CLINICAL TRIAL: NCT02215902
Title: A Clinical Safety Study of the Aethlon Hemopurifier® in Chronic ESRD Patients With HCV Infection
Brief Title: Safety Study of the Aethlon Hemopurifier
Acronym: AEMD-IDE-20
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Adequate safety data has been accumulated and the # of patients meeting inclusion criteria has diminished.
Sponsor: Aethlon Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEMD - IDE - 2013
Record Dates: First submitted 2014-08-12; First posted 2014-08-13 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: End Stage Renal Disease; Hepatitis C Infection
Keywords: ESRD; Hepatitis C
MeSH Terms: conditions — Kidney Failure, Chronic; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hemopurifier (Experimental): Affinity plasmapheresis
  Interventions: Device: Affinity plasmapheresis

INTERVENTIONS:
Device: Affinity plasmapheresis — Insert investigational affinity plasma filter into hemodialysis circuit during routine hemodialysis treatments.
  Other Names: Aethlon Medical Hemopurifier

SUMMARY:
Primary Objectives:

To demonstrate the safety of the Aethlon Hemopurifier® when used in extracorporeal blood purification.

Secondary Objectives:

To quantify the number of viral copies captured by the Aethlon Hemopurifier® during the first and last Hemopurifier treatments using elution methods developed by Aethlon Medical Inc.

To measure changes in viral load in patients before and after treatment with the Aethlon Hemopurifier®.

DETAILED DESCRIPTION:
This will be a single-arm, sequential, controlled feasibility/safety study in which each subject will serve as his/her own control. The control period will be the week immediately preceding the use of the investigational device during which eligible subjects will undergo and be monitored during three standard intermittent dialysis sessions. Vital signs, blood chemistries, hematology, liver function and adverse events will be measured. On weeks two and three, patients will receive treatment with the Hemopurifier® three times per week coincident with their ongoing standard intermittent hemodialysis treatments. During these two weeks, subjects will be assessed for the same clinical parameters but with the addition of viral load determination by quantitative PCR before and after each treatment with the Hemopurifier®. Viral load will also be measured at follow-up prior to the start of a given subject's hemodialysis treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 18 years of age and older.
2. Positive test for HCV infection (any genotype).
3. End-stage-renal disease (ESRD) requiring dialysis - already established on HD.
4. The arteriovenous fistula, graft or central venous catheter must have been functioning adequately for at least 1 month before entry into study showing no signs of infection or blockage.
5. Have recovered from the toxicity of any prior systemic therapy.
6. Ability to tolerate blood volume losses of up to 150 ml per week, i.e. 50 ml each.
7. Stable clinical condition, including stable hemoglobin which has not fluctuated more than 1.5 -2.0 gm/dl within 28 days prior to enrollment into study.
8. Must have the following minimum hematologic, biochemical, and serologic criteria documented within 28 days prior to enrollment into study:

   1. Hemoglobin values of ≥ 9.5 gm/dL for males and females
   2. Platelet count > 100,000/mm3
   3. Bilirubin < 4 mg/dL
   4. Albumin stable and not less than 3.5 g/dl.
9. Women of child-bearing potential must be practicing barrier or oral contraception for the duration of the study or documented as surgically sterile or one year post-menopausal.
10. If female, be non-nursing, non-pregnant and have a negative serum or urine pregnancy test within two weeks of starting study.
11. The subject must be informed of the investigational nature of this study and written informed consent obtained prior to enrollment in this study.
12. The subject must be able to comprehend the study description and its nature as only a feasibility study.

Exclusion Criteria:

1. Administration of Pegasys-ribavirin or ANY anti-viral drug therapy within 90 days prior to enrollment into study.
2. Administration of any other investigational drugs within 90 days prior to enrollment into study.
3. Clinically significant infection, other than HCV, defined as any acute or chronic viral, bacterial, or fungal infection, which requires specific therapy (Anti-infectious therapy must have been completed at least 14-days before entry into study) in order to make entry into the study possible.
4. Patient infected with human immunodeficiency virus or has AIDS.
5. A history of hypotensive episodes during dialysis which lead to early termination of the treatment in the 2 treatments prior to the start of study treatments.
6. Patients who have received an ACE (angiotensin converting enzyme) inhibitor within the last 24 hours should not be treated. Patients receiving an ACE inhibitor may experience an anaphylactoid-like reaction, including hypotension associated with flushing, dyspnea, and bradycardia. Such reactions, if left untreated, may be life-threatening. The administration of ACE inhibitors also has been associated with the occurrence of tachycardia. Risk of an anaphylactoid-like reaction or tachycardia may be minimized by the temporary cessation of the administration of ACE inhibitors for 6 days or longer before initiating the treatment protocol.
7. Any known pre-existing medical condition that could interfere with the subject's participation in the entire protocol, including serious psychiatric disorders, CNS trauma or active seizure disorders requiring medication, poorly-controlled diabetes mellitus as indicated by an Hb-A1c > 8% within the two weeks prior to protocol initiation, significant cardiovascular dysfunction within the past 6 months (e.g., angina, congestive heart failure, recent myocardial infarction, severe interdialytic hypotension, or significant arrhythmia).
8. Subjects with ECG showing clinically significant abnormalities.
9. Dementia or other cognitively-limiting disease processes which would make it difficult for the patient to articulate their clinical status.
10. Prior blood transfusion for any reason within 3 months prior to enrollment into study.
11. Recent history of bleeding or bleeding disorders that would likely require the restriction in use of heparin during study treatments.
12. Active immunologically mediated disease (e.g., inflammatory bowel disease [Crohn's disease, ulcerative colitis], rheumatoid arthritis, idiopathic thrombocytopenia purpura, systemic lupus erythematosus, autoimmune or inherited hemolytic anemia, scleroderma, severe psoriasis).
13. Any medical condition requiring, or likely to require during the course of the study, chronic systemic administration of steroids or other immunoregulatory medications.
14. Substance abuse, such as alcohol (~80 gm/day), IV drugs, and inhaled drugs (If the subject has a history of substance abuse, to be considered for inclusion into the protocol, the subject must have abstained from using the abused substance for at least 2 months. Subjects receiving methadone within the past year are also excluded.)
15. Any cancer requiring systemic chemotherapy or radiotherapy.
16. Any other condition that, in the opinion of the Principal Investigators, would make the subject unsuitable for enrollment, or could interfere with the subject participating in and completing the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-12; Primary Completion 2017-03-10 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
Rate of adverse events | 30 days

SECONDARY OUTCOMES:
Viral load reduction | 2 weeks
  Viral load will be measured before and after each treatment with the investigational device.

OTHER OUTCOMES:
Quantification of viral copies captured. | 2 weeks
  The number of viral copies captured by the Aethlon Hemopurifier® during the first and last Hemopurifier treatments will be quantified.

CONTACTS AND LOCATIONS:
Overall Officials: Felicia B Ricks, RD CS-R LD, Study Director — DaVita Clincal Research; Ronald Ralph, M. D. FASN, Principal Investigator — Kidney Associates, PLLC
Locations (1):
- DaVita Med Center Dialysis, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided